CLINICAL TRIAL: NCT03304210
Title: Intraperitoneal Aerosolization of Albumin-stabilized Paclitaxel Nanoparticles for Stomach, Pancreas, Breast and Ovarian Cancer
Brief Title: PIPAC Nab-pac for Stomach, Pancreas, Breast and Ovarian Cancer
Acronym: PIPAC-nabpac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other); University Ghent (Other); Hopital Lariboisière (Other); University Women's Hospital Tübingen (Other); Candiolo Cancer Institute - IRCCS (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AGO/2017/003
Record Dates: First submitted 2017-09-11; First posted 2017-10-06 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Peritoneal Carcinomatosis; Ovarian Cancer Stage IIIB; Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV; Breast Cancer Stage IIIB; Breast Cancer Stage IIIc; Breast Cancer Stage IV; Stomach Cancer Stage III; Stomach Cancer Stage IV With Metastases; Pancreas Cancer, Stage III; Pancreas Cancer, Stage IV
Keywords: PIPAC; Peritoneal carcinomatosis; Ovarian cancer; Pharmacokinetics; Pharmacodynamics; Safety and efficacy; Abraxane; Breast cancer; Pancreas cancer; Stomach cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Abraxane 35 mg/m² (Experimental): PIPAC with Abraxane (35 mg/m²) will be administered every 4 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Abraxane
- Abraxane 70 mg/m² (Experimental): PIPAC with Abraxane (70 mg/m²) will be administered every 4 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Abraxane
- Abraxane 90 mg/m² (Experimental): PIPAC with Abraxane (90 mg/m²) will be administered every 4 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Abraxane
- Abraxane 112.5 mg/m² (Experimental): PIPAC with Abraxane (112.5 mg/m²) will be administered every 4 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Abraxane
- Abraxane 140 mg/m² (Experimental): PIPAC with Abraxane (140 mg/m²) will be administered every 4 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Abraxane

INTERVENTIONS:
Drug: PIPAC with Abraxane — Albumin bound nanoparticle paclitaxel (Abraxane) will be administered intraperitoneally using the PIPAC technique. The administered dose will escalate ranging from 35 to 140 mg/m². PIPAC will be performed every 4 weeks for 3 cycles.

SUMMARY:
The PIPAC nab-pac study is designed to examine the maximal tolerated dose of albumin bound nanoparticle paclitaxel (nab-pac, Abraxane) administered with repeated pressurized intraperitoneal aerosol chemotherapy (PIPAC), in a multicentre, multinational phase I trial.

DETAILED DESCRIPTION:
Over 85% of women with ovarian cancer (OC) will develop a peritoneal recurrence after initial therapy. The prognosis of patients with recurrent disease is poor, with a median survival ranging from 12 to 24 months. Most of these patients ultimately develop platinum resistant disease (PROC). Current systemic therapy results in a very modest improvement of progression free and overall survival. The addition of locoregional, intraperitoneal (IP) therapy may improve disease control in recurrent OC. Recently, pressurized intraperitoneal aerosol therapy (PIPAC) was added to the therapeutic arsenal. This novel technique allows repeated laparoscopy aided aerosol delivery of anticancer drugs to the peritoneal cavity. Abraxane (nab-pac, Celgene) is a novel 130 nm, albumin-bound (nab) nanoparticle formulation of paclitaxel which has noteworthy single-agent activity and a favourable toxicity profile when used systemically in PROC. A recent phase I study showed a significant pharmacokinetic advantage after IP instillation of nab-pac in patients with peritoneal carcinomatosis from ovarian or gastro-intestinal (GI) origin.

In phase I of this study, dose escalation will be combined with pharmacokinetic/pharmacodynamic modelling which incorporates, in addition to plasma, tumour tissue, and peritoneal drug concentrations, biomarkers of toxicity and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Phase I study: patients with advanced carcinomatosis from ovarian, breast, gastric, or pancreatic origin. No alternative systemic treatment options are available.
* Age over 18 years
* Adequate performance status (Karnofsky index > 60%)
* Absence of intestinal or urinary obstruction
* Limited size of the majority of peritoneal tumor implants (< 5 mm)
* Absent or limited ascites
* Ability to understand the proposed treatment protocol and provide informed consent
* Expected life expectancy more than 6 months
* Laboratory data

  * Serum creatinine ≤ 1.5 mg/dl or a calculated GFR (CKD-EPI) ≥ 60 mL/min/1.73 m²
  * Serum total bilirubin ≤ 1.5 mg/dl, except for known Gilbert's disease
  * Platelet count > 100.000/µl
  * Hemoglobin > 9g/dl
  * Neutrophil granulocytes > 1.500/ml
  * No major blood coagulation disorders. Parameters within normal range.
* Absence of alcohol and/or drug abuse
* No other concurrent malignant disease
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding. Women who can become pregnant must ensure effective contraception.
* Active bacterial, viral or fungal infection
* Active gastro-duodenal ulcer
* Parenchymal liver disease (any stage cirrhosis)
* Uncontrolled diabetes mellitus
* Psychiatric pathology affecting comprehension and judgement faculty
* General or local (abdominal) contra-indications for laparoscopic surgery
* Documented intolerance or allergy to paclitaxel
* Patients who receive other taxane therapy until three weeks before the first experimental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wim P Ceelen, MD, PhD, Prof, Principal Investigator — University Hospital, Ghent
Locations (1):
- UZ Ghent, Ghent, East-Flanders, Belgium

REFERENCES:
- [Background] Van De Sande L, Graversen M, Hubner M, Pocard M, Reymond M, Vaira M, Cosyns S, Willaert W, Ceelen W. Intraperitoneal aerosolization of albumin-stabilized paclitaxel nanoparticles (Abraxane) for peritoneal carcinomatosis - a phase I first-in-human study. Pleura Peritoneum. 2018 Jun 8;3(2):20180112. doi: 10.1515/pp-2018-0112. eCollection 2018 Jun 1. PMID 30911657
- [Result] Ceelen W, Sandra L, de Sande LV, Graversen M, Mortensen MB, Vermeulen A, Gasthuys E, Reynders D, Cosyns S, Hoorens A, Willaert W. Phase I study of intraperitoneal aerosolized nanoparticle albumin based paclitaxel (NAB-PTX) for unresectable peritoneal metastases. EBioMedicine. 2022 Aug;82:104151. doi: 10.1016/j.ebiom.2022.104151. Epub 2022 Jul 15. PMID 35843174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Started | 2 | 2 | 3 | 3 | 10
Completed | 2 | 2 | 3 | 3 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m² | Total
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 3 | 2 | 9 | 15
  >=65 years | 1 | 2 | 0 | 1 | 1 | 5
Age, Continuous [Median (Full Range); unit: years] | 64 [62 to 65] | 68 [67 to 68] | 52 [49 to 58] | 59 [47 to 70] | 51 [28 to 66] | 57 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 7 | 12
  Male | 1 | 0 | 3 | 1 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) of Abraxane
Description: The MTD was defined as the highest dose of aerosolized Abraxane, administered 3 times using PIPAC, that does not cause unacceptable side effects. Dose limiting toxicity was recorded in a 14 week-window starting from the first PIPAC and defined a priori as any of the following: 1. any Grade 3 or 4 non-hematologic toxicity excluding fatigue and controllable nausea, vomiting, abdominal pain, and diarrhoea; 2. grade 4 thrombocytopenia; 3. grade 4 neutropenia lasting more than 7 days or associated with fever; 4. failure to perform more than one PIPAC due to toxicity; 5. surgical complication Dindo-Clavien grade IIIB or higher.
  In order to optimize the balance between safety and efficacy, we used a time-to-event continual reassessment model (TITE-CRM), where an initial design was followed until the first DLT occurred. Conservative a priori estimates of DLT were used to calculate the original dose escalation scheme.
Time Frame: Within 14 weeks of the start of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Surgical Morbidity
Description: Surgical complications were scored using the Clavien Dindo classification. Grade I: Any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention. This includes the need for certain drugs (e.g. antiemetics, antipyretics, analgesics, diuretics and electrolytes), treatment with physiotherapy and wound infections that are opened at the bedside Grade II: Complications requiring drug treatments other than those allowed for Grade I complications; this includes blood transfusion and total parenteral nutrition (TPN) Grade III: Complications requiring surgical, endoscopic or radiological intervention Grade IV: Life-threatening complications; this includes CNS complications (e.g. brain haemorrhage, ischaemic stroke, subarachnoid haemorrhage) which require intensive care, but excludes transient ischaemic attacks (TIAs) Grade V: Death of the patient
Time Frame: 6 months after third PIPAC
Measure: Number; unit: participants
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
participants | 2 | 2 | 3 | 3 | 10

3. Secondary Outcome: Maximum Plasma Concentration of Abraxane
Description: Abraxane will be measured in plasma, using UPLC-MS/MS.
Time Frame: T = 0 minutes, T = 15 minutes, T = 30 minutes, T = 60 minutes, T = 1.5 hour, T = 2 hours, T = 4 hours, T = 8 hours, T = 12 hours, T = 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
ng/mL | 58 (15) | 138 (42) | 101 (13) | 157 (49) | 184 (68)

4. Secondary Outcome: Area Under The Curve (AUC) of Abraxane
Description: Abraxane will be measured in plasma, using LC-MS/MS.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
h*ng/mL | 585 (93) | 962 (237) | 813 (99) | 1658 (465) | 2002 (569)

5. Secondary Outcome: Histological Response Via Peritoneal Regression Grading Scoring (PRGS)
Description: Punch biopsies are taken at the same location, which are marked with a stainless-steel surgical clip during each PIPAC procedure. Samples are fixed in 4% paraformaldehyde in PBS for 72 hours and embedded in paraffin. Tissues are serially sectioned and stained with haematoxylin & eosin; immunohistochemical staining is performed for epithelial cellular adhesion molecule (EpCAM). The peritoneal regression grading score (PRGS) is determined by a GI pathologist.
  The mean score of all samples is calculated per treatment, and percentage changes in mean PRGS between successive PIPAC treatments is calculated. The unit of measure represented is the amount of participants in which tumor regression was observed.
Time Frame: T = 0 minutes, before nebulization
Population: Tumour tissue samples were taken from each abdominal quadrant (n = 4) before aerosol delivery. In 30% of all procedures, less than four biopsies (or none) were taken due to technical reasons (adhesions) or because no visible tumour was present, which explains the lower number of participants analyzed.
Measure: Number; unit: participants with tumor regression
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 8
participants with tumor regression | 0 | 1 | 1 | 0 | 7

6. Secondary Outcome: Neutropenia - Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Blood samples will be collected to analyse the absolute neutrophil count
Time Frame: Pre-operatively, and 12 hours, 24 hours and 1 week after each PIPAC
Measure: Count of Participants; unit: Participants
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
Participants
  CTCAE grade <=2 | 0 | 0 | 1 | 1 | 4
  CTCAE grade >2 | 0 | 0 | 0 | 0 | 1
  no neutropenia | 2 | 2 | 2 | 2 | 5

7. Secondary Outcome: Decreased Platelets - Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Blood samples will be collected to analyse the amount of platelets.
Time Frame: Pre-operatively, and 12 hours, 24 hours and 1 week after each PIPAC
Measure: Count of Participants; unit: Participants
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
Participants
  CTCAE grade <=2 | 0 | 1 | 1 | 2 | 3
  CTCAE grade >2 | 0 | 0 | 1 | 0 | 0
  no thrombopenia | 2 | 1 | 1 | 1 | 7

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Abraxane 35 mg/m² | Abraxane 70 mg/m² | Abraxane 90 mg/m² | Abraxane 112.5 mg/m² | Abraxane 140 mg/m²
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/2 | 1/3 | 1/3 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/3 | 1/3 | 6/10
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abraxane 35 mg/m² (N=2) | Abraxane 70 mg/m² (N=2) | Abraxane 90 mg/m² (N=3) | Abraxane 112.5 mg/m² (N=3) | Abraxane 140 mg/m² (N=10)
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intestine obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
thrombocytopenia grade 3 (CTCAE) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
progression peritoneal disease leading to death (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
surgical wound infection (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
anaphylactic shock during surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
infection peritoneum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anorexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abraxane 35 mg/m² (N=2) | Abraxane 70 mg/m² (N=2) | Abraxane 90 mg/m² (N=3) | Abraxane 112.5 mg/m² (N=3) | Abraxane 140 mg/m² (N=10)
thrombopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
white blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 9 (9)
elevated AST (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 6 (6)
elevated ALT (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 4 (4)
elevated ALP (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
elevated bilirubin (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
elevated GGT (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 7 (7)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
bleeding at incision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
paralytic ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (7)
electrocardiogram T wave abnormal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bacterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
surgical wound infection (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
edema lower limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
allergic reaction to anesthesia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03304210/Prot_SAP_000.pdf